CLINICAL TRIAL: NCT00402012
Title: Pioglitazone Reverses Defects in Mitochondrial Biogenesis in Patients With T2DM
Brief Title: "TAKE TIME" Pioglitazone Reverses Defects in Mitochondrial Biogenesis in Patients With T2DM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Principal Investigator, Frank Greenway, Clinical Medical Doctor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PBRC 26027
Record Dates: First submitted 2006-11-17; First posted 2006-11-22 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention)
- 2 (Experimental)
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — During the double-blind, 12 weeks treatment period, subjects will self-administer study medication (pioglitazone or equivalent volume of placebo) 30 mg/day each morning. The dose of pioglitazone will be increased to 45 mg/day after 4 weeks if the fasting plasma glucose is higher than 100mg/dl or the HbA1C is higher than 7%. This dose has proven tolerability, safety and efficacy for type 2 diabetes and has previously been used at the Pennington Center in studies on pioglitazone.
  Other Names: TZD
  Arms: 2

SUMMARY:
This study is designed to look at the effect of Pioglitazone treatment on the body's ability to burn food in order to produce energy.

DETAILED DESCRIPTION:
Skeletal muscle mitochondrial defects are a sine qua non of insulin resistance in patients with T2DM. Pioglitazone decreases free fatty acid levels and restores mitochondria number in adipose tissue whereas high fat diet and lipid infusion decreases genes involved in mitochondrial biogenesis. Increased lipid flux from diet or adipose tissue into skeletal muscle might be the cause of decreased mitochondrial biogenesis. The purpose of this study is to determine if 22 weeks treatment with Pioglitazone can increase mitochondrial biogenesis in muscle in 30 uncomplicated T2DM patients that were previously not taking TZD's. This Phase IV, randomized, double-blind, placebo controlled, clinical trial will consist of 3 phases: a screening, a placebo / Pioglitazone phase (12 weeks) and a weight loss period (6-10 weeks). The primary endpoint is to identify the changes in skeletal muscle mitochondria number and gene expression. Secondary endpoints include MRS measured mitochondrial capacity, insulin sensitivity for glucose disposal and insulin suppression of free fatty acids, electron transport chain activity, mitochondrial content and intra hepatic and intra myocellular lipid. Metformin and Sulfonylurea will be used as standardized oral therapy to maintain HbA1C < 7.0. After completing the protocol, patients will be offered a very low calorie liquid diet (800kcal/d) to assist them in losing weight. During this period they will continue on their previously randomized treatment. When patients lose 10% of their body weight, patients will be switched to a weight maintenance diet (meal replacement with 1 can of glucerna at breakfast and lunch with a "healthy" dinner) for 10 days. MRS measured mitochondrial capacity will again be determined to see if weight loss + pioglitazone has more effect on mitochondrial function than pioglitazone alone.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-70 with Type 2 diabetes as defined by:

  * Fasting plasma glucose > 126 mg/dL at entry
  * Or a two-hour OGTT glucose > 200mg/dL
  * Or current treatment with one or two oral anti-diabetic drugs, except TZD
  * Or currently using insulin
* Fasting plasma glucose < 200mg/dL at entry
* BMI >27.0 and <45.0kg/m2
* Adequate contraception for women (including, but not limited to: oral contraception, hysterectomy, tubal ligation, or post-menopausal as defined by > 6 months without a menstrual cycle and FSH > 40 mIU/ml).

Exclusion Criteria:

* Significant renal, cardiac, liver, lung, or neurological disease (controlled hypertension is acceptable if baseline bp < 140/90 on medications).
* Prior use of other thiazolidinediones (rosiglitazone [AVANDIATM], pioglitazone [ACTOSTM])
* Use of drugs known to affect energy metabolism or body weight: including, but not limited to: orlistat, sibutramine, ephedrine, phenylpropanolamine, corticosterone, etc.
* Pregnancy
* Alcohol or other drug abuse
* Unwilling or unable to abstain from caffeine (48h) and tobacco (24h) prior to metabolic rate measurements
* Increased liver function tests at baseline (AST/ALT/GGT/or alkaline phosphatase greater than 2.5 times the upper limit of normal)
* Metal objects that would interfere with the measurement of body composition /MRS such as implanted rods, surgical clips, etc.
* HbA1C of > 10%.
* NYHA class III/IV CHF is an exclusionary cardiac condition.
* history of deep vein thrombosis (DVT) or pulmonary embolism (PE)
* varicose veins
* major surgery on the abdomen, pelvis, or lower extremities within previous 3 months
* cancer (active malignancy with or without concurrent chemotherapy)
* rheumatoid disease
* bypass graft in limb
* known genetic factor (Factor V Leiden, etc) or hypercoagulable state
* diagnosed peripheral arterial or vascular disease, or intermittent claudication
* family history of primary DVT or PE (pulmonary embolism)
* peripheral neuropathy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-11; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Change in skeletal muscle mitochondrial number (electron microscopy + qPCR of mtDNA) and mitochondrial gene expression in T2DM patients treated with pioglitazone (vs. placebo) | baseline and after intervention

SECONDARY OUTCOMES:
insulin sensitivity for insulin suppression of free fatty acid and glucose disposal | baseline and after intervention
electron transport chain activity; mitochondrial content by MRS (ATP max) | baseline and after intervention
intra hepatic and intra myocellular lipid by MRS; mitochondrial content by MRS (ATP max) post weight loss period | baseline ,after treatment and after weight loss

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Smith, M.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Bajpeyi S, Myrland CK, Covington JD, Obanda D, Cefalu WT, Smith SR, Rustan AC, Ravussin E. Lipid in skeletal muscle myotubes is associated to the donors' insulin sensitivity and physical activity phenotypes. Obesity (Silver Spring). 2014 Feb;22(2):426-34. doi: 10.1002/oby.20556. Epub 2013 Sep 10. PMID 23818429
- [Derived] Bajpeyi S, Pasarica M, Moro C, Conley K, Jubrias S, Sereda O, Burk DH, Zhang Z, Gupta A, Kjems L, Smith SR. Skeletal muscle mitochondrial capacity and insulin resistance in type 2 diabetes. J Clin Endocrinol Metab. 2011 Apr;96(4):1160-8. doi: 10.1210/jc.2010-1621. Epub 2011 Feb 9. PMID 21307136
- [Derived] Costford SR, Bajpeyi S, Pasarica M, Albarado DC, Thomas SC, Xie H, Church TS, Jubrias SA, Conley KE, Smith SR. Skeletal muscle NAMPT is induced by exercise in humans. Am J Physiol Endocrinol Metab. 2010 Jan;298(1):E117-26. doi: 10.1152/ajpendo.00318.2009. Epub 2009 Nov 3. PMID 19887595